CLINICAL TRIAL: NCT04903379
Title: An Evaluation of an Online Webinar Aimed at Shifting the Beliefs of the UK Population Regarding Persistent Pain
Brief Title: Flippin Pain: A Public Health Campaign Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Teesside University (Other)
Collaborators: Prof Denis Martin (Unknown); Prof Cormac Ryan (Unknown); Gail Sowden (Unknown)
Responsible Party: Principal Investigator, Nick Livadas, Mr Nick Livadas, Teesside University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6167
Record Dates: First submitted 2021-05-23; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Pain, Chronic
Keywords: Education
MeSH Terms: conditions — Chronic Pain | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: All webinar registrants will be invited to participate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain science education and self management strategies (Other): The intervention will be educational in the form of the provision of contemporary pain science education and supportive advice from people with a history of persistent pain. The duration of the webinar will be 90 minutes.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — An explanation of contemporary pain science and a description of effective treatment strategies used by people with a history of persistent pain.

SUMMARY:
An online webinar aiming to improve the public beliefs related to persistent pain will be offered to members of the public in the UK via social media and targeted via written invitation to individuals on a waiting list for pain and musculoskeletal services in Ayrshire and Arran, Scotland.

DETAILED DESCRIPTION:
Flippin Pain is a UK based public health campaign which aims to shift the populations perception related to persistent pain to one that is aligned with contemporary pain science understanding. The webinar will be presented by a panel consisting of people with a history of persistent pain and healthcare professionals with experience of treating persistent pain. The webinar will be advertised on social media. When registrants receive their confirmation email confirming their place they will be notified of of the invitation to participate. This link within the email will take them to an online participant information sheet. Once this is read they may decide to proceed with an online survey which would take 10 minutes to complete. This survey will include some non identifiable demographic data and the Pain Beliefs Questionnaire (PBQ). The PBQ is a validated tool that does not require a license to use. The survey will be administered immediately after the webinar, at 3, 6 and 12 months to assess for longitudinal changes in pain beliefs. Another recruitment strategy will be the posted invitation to individuals on a National health Service waiting list. Both groups will complete the same survey questions. The last question of the survey will request the participants email so that future surveys can be sent and the follow ups linked by participant. Individuals will also be asked within the survey if they consent to further contact about the opportunity to answer questions vie a telephone/online interview related to their experience of the webinar. Purposive sampling will be used to recruit 15-20 individuals for a semi structured interview.

ELIGIBILITY:
Inclusion Criteria:

* Resident within the United Kingdom
* Over the age of 18 years

Exclusion Criteria:

* Unable to read the English version of the surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Beliefs Questionnaire | 10 minutes to complete
  A validated self reported questionnaire
Pain self efficacy questionnaire | 10 minutes to complete
  A validated self reported questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ayrshire and Arran NHS Scotland, Kilmarnock, Ayrshire and Arran, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Non identifiable data may be shared.